CLINICAL TRIAL: NCT00855179
Title: A 12-week, Double-blind, Randomised, Placebo-controlled, Multicentre Trial to Evaluate Efficacy and Tolerability of Antistax® Film Coated Tablets, 720 mg/Day Orally, in Male and Female Patients Suffering From Chronic Venous Insufficiency
Brief Title: Assess the Efficacy and Tolerability of Antistax Film-coated Tablets in Patients With Chronic Venous Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1138.11
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency | interventions — AS 195

ARMS (2):
- Antistax film-coated tablets 360 mg (Active Comparator): Patient to receive 2 tablets daily as a morning dose, each containing 360 mg Antistax
  Interventions: Drug: Red vine leaf extract (AS 195)
- Placebo (Placebo Comparator): Patient to receive 2 tablets identical to those containing 360 mg Antistax daily as a morning dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Red vine leaf extract (AS 195) — Antistax film-coated tablet 360 mg
  Arms: Antistax film-coated tablets 360 mg
Drug: Placebo — Placebo tablets identical to those containing Anstistax 360 mg
  Arms: Placebo

SUMMARY:
To assess the efficacy and tolerability of Antistax film coated tablets in patients with chronic venous insufficiency (CVI, CEAP Classification: Clinical class 3 and 4a).

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. 18 years of age or older
3. CVI, Clinical Class 3 and Class 4a according to the CEAP classification
4. Presence of stable edema determined by a pretibial pit after 30 seconds pressure with the thumb documented by a photo
5. Stable and reproducible status of swelling documented by difference of less than 150g between screening and baseline as determined by water displacement method
6. Presence of moderate to severe varicoses (dilated, tortuous veins in the subcutaneous tissue with a diameter of more than 3mm
7. Intensity of leg pain at least 5 cm on the Visual Analogue Scale at baseline and presence of hyperpigmentation or eczema and presence of moderate to severe edema
8. Willing and able to give written informed consent prior to participation in the trial
9. Patients expected to be compliant (compliance with run-in medication greater than 80% as checked by drug count)

Exclusion Criteria:

1. Decompensated cardiac insufficiency according to the New York Heart Association (NYHA) classification III and IV for cardiac patients
2. Edema not due to venous disease of the legs(e.g. latent cardiac insufficiency, renal insufficiency, lymphoedema, etc)
3. Severe skin changes, e.g. lipodermatosclerosis
4. Current florid venous ulcer
5. Peripheral arterial disease (ankle/arm pressure index less than 0.9)
6. Untreated or insufficiently controlled hypertension
7. Current acute phlebitis of thrombosis with the last 3 months. Post-thrombotic syndrome, who do not currently receive an anticoagulation treatment can be included in the trial
8. Renal insufficiency
9. Liver disease; hepatic insufficiency
10. Hyper- or hypocalcemia
11. Malignancies
12. Anamnestic indications of diabetic microangiopathy or polyneuropathy
13. Drug and/or alcohol abuse
14. Severe climacteric complaints; changes in or initiation of post-menopausal hormone replacement therapy within the last 3 months
15. Immobility
16. Avalvulia
17. Klippel-Trénaunay-Weber-Syndrome
18. State after pulmonary embolism
19. Recognized hypersensitivity to the trial drug ingredients
20. Clinical indication for a specific phlebologic treatment, e.g. compression treatment phlebectomy, etc

Previous Treatments:

1. Compression therapy and/or wearing of support stockings less than 2 weeks prior to the visit at baseline
2. Venous surgery or sclerotherapy with the last 3 months at the leg used for volumetry
3. Treatment with drugs affecting the veins less than 4 weeks prior to visit 1
4. Changes in or unstable response to treatment with theophylline, cardiac glycosides, ACE-inhibitors, calcium antagonists, or laxatives with the last 2 weeks prior to visit 1

Concomitant Treatment:

1. Compression therapy
2. Diuretics
3. Nitrates
4. Ergot alkaloids
5. All preparations which are used as compounds for venous therapy in CVI (e.g. vasoprotectives for antivaricose therapy, preparations with heparin, sclerosing agents, flavonoid-containing preparations, other phytopharmaceuticals
6. Other drugs active on blood vessels and circulation
7. Extensive use of laxatives
8. Anticipated changes in the intake of hormones, ie contraceptives
9. Scheduled major surgery requiring full anesthesia

Other exclusion Criteria:

1. Previously studied under the present protocol
2. Participation in another clinical trial within less than 90 days prior to Visit 1
3. Participation in another clinical trial during the present trial
4. Patient is investigator, co-investigator, trial nurse in this trial or is a relative of the investigator, co-investigator or trial nurse in this trial
5. Pregnant or nursing women or inadequate birth control methods (this applies to females of childbearing potential only; reliable contraceptive methods are hormonal contraceptives, intrauterine devices, sexual abstinence of sterilization)
6. Patients considered as mentally ill as well as unable to work or with limited working ability, or unable (or only partially able) to follow the spoken or written explanations concerning the trial
7. Patients in bad general health state according to the investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in limb volume determination at day 84 (water displacement method) | 84 days

SECONDARY OUTCOMES:
Change from baseline in limb volume determination at day 21 and 42 (water displacement method) | 21 and 42 days
Change from baseline in the subjective symptoms of CVI (tired, heavy legs, sensation of tension in the legs) pain in the legs) measured by Visual Analogue Scales at day 21,42 and 84 | 21, 42 and 84 days
Incidence of adverse events | 84 days
Global assessment of efficacy by the patient at day 84 | 84 days
Change from baseline in the calf circumference at day 21, 42 and 84 | 21, 42 and 84 days
Global assessment of efficacy by the investigator at day 84 | 84 days
Time to improvement in symptoms | 84 days
Vital signs (pulse rate, blood pressure) | 84 days
Number of patients with abnormal Serum Laboratory Parameters | 84 days
Global assessment of tolerability by the patient at day 84 | 84 days
Global assessment of tolerability by the investigator at day 84 | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (20):
- Germany (20):
  - 1138.11.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 1138.11.49016 Boehringer Ingelheim Investigational Site, Berlin
  - 1138.11.49019 Boehringer Ingelheim Investigational Site, Bochum
  - 1138.11.49014 Boehringer Ingelheim Investigational Site, Bonn
  - 1138.11.49023 Boehringer Ingelheim Investigational Site, Breisach
  - 1138.11.49003 Boehringer Ingelheim Investigational Site, Coburg
  - 1138.11.49013 Boehringer Ingelheim Investigational Site, Cologne
  - 1138.11.49024 Boehringer Ingelheim Investigational Site, Dülmen
  - 1138.11.49007 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1138.11.49020 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1138.11.49009 Boehringer Ingelheim Investigational Site, Greifswald
  - 1138.11.49010 Boehringer Ingelheim Investigational Site, Lübeck
  - 1138.11.49011 Boehringer Ingelheim Investigational Site, Mainz
  - 1138.11.49012 Boehringer Ingelheim Investigational Site, Minden
  - 1138.11.49005 Boehringer Ingelheim Investigational Site, München
  - 1138.11.49022 Boehringer Ingelheim Investigational Site, Oberhausen
  - 1138.11.49002 Boehringer Ingelheim Investigational Site, Oberkirch
  - 1138.11.49001 Boehringer Ingelheim Investigational Site, Rottach-Egern
  - 1138.11.49006 Boehringer Ingelheim Investigational Site, Rottweil
  - 1138.11.49018 Boehringer Ingelheim Investigational Site, Tübingen

REFERENCES:
- [Derived] Rabe E, Stucker M, Esperester A, Schafer E, Ottillinger B. Efficacy and tolerability of a red-vine-leaf extract in patients suffering from chronic venous insufficiency--results of a double-blind placebo-controlled study. Eur J Vasc Endovasc Surg. 2011 Apr;41(4):540-7. doi: 10.1016/j.ejvs.2010.12.003. Epub 2011 Jan 15. PMID 21239190